CLINICAL TRIAL: NCT01151254
Title: Comparison of Propofol Based Anesthesia and Postoperative Sedation (PA) Versus Volatile Anesthetics Based Anesthesia and Postoperative Sedation (VA) in Cardiac Surgical Patients
Brief Title: Comparison of Propofol Based Versus Volatile Based Anesthesia and Postoperative Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHN REB 06-0159 B
Record Dates: First submitted 2010-05-17; First posted 2010-06-28 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Cardiac Surgery
Keywords: Cardiac Surgery; Sedation; Intensive care; Volatile anesthesia; Intravenous anesthesia; Pre and post conditioning after cardiac surgery
MeSH Terms: interventions — Isoflurane; Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA-Intravenous Sedation (Active Comparator): Propofol based total intravenous anesthesia and postoperative sedation
  Interventions: Other: Propofol
- Volatile sedation (Active Comparator): Total inhalational anesthesia and postoperative sedation with the AnaConda device
  Interventions: Drug: Isoflurane/sevoflurane

INTERVENTIONS:
Drug: Isoflurane/sevoflurane — Volatile for sedation in the CVICU while intubated
  Other Names: 2-chloro-2-(difluoromethoxy)-1,1,1-trifluoro-ethane; 2,2,2-trifluoro-1-[trifluoromethyl]ethyl fluoromethyl ether
  Arms: Volatile sedation
Other: Propofol — Propofol for sedation in the CVICU
  Other Names: Diprivan
  Arms: PA-Intravenous Sedation

SUMMARY:
All patients undergoing cardiac surgery require intraoperative anesthesia and short-term postoperative sedation with anesthetic agents after the procedure when patient is in the intensive care unit (ICU). The clinical data obtained so far are concentrating on intraoperative use volatile agents (preconditioning) resulting in better postoperative cardiac function and less release of biochemical markers of myocardial damage. There are no studies investigating whether postoperative use of volatile agents (post conditioning) in cardiac surgical population is improving outcomes. The aim of the present study is to compare total intravenous anesthesia and postoperative sedation versus total volatile anesthesia and postoperative sedation in cardiac surgical population.

ELIGIBILITY:
Inclusion criteria:

* Patients scheduled for coronary artery bypass graft surgery with good ventricular function (grade 1-2 ventricle)
* Signed informed consent

Exclusion criteria:

* Patients undergoing valvular surgery
* Severe kidney or liver disease (creatinine > 2.5mg.dL-1 and bilirubin > 2 mg.dL-1)
* Patients with known hypersensitivity to any of the trial drugs (propofol, volatile anesthetics), e.g. propofol allergy or malignant hyperthermia (induced by volatile anesthetics)
* Patient with poorly controlled diabetes or on oral anti-diabetic medication (inhibit preconditioning caused by volatile anesthetics)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The composite primary end point of the trial will be the development of enzymatic signs of myocardial injury or MI, postoperative low output syndrome, or both. Enzymatic MI will be determined after obtaining serial measurements of troponin. | Measurements of troponin levels will be after induction of anesthesia (baseline) and at 0, 2, 4, 8, and 24 h after arrival into the ICU.

SECONDARY OUTCOMES:
Quality of sedation | Post ICU arrival POD 0 to discharge (2hours to on average 5-7 days until discharge)
Incidence of delirium | Post ICU arrival POD 0 to discharge (2hours to on average 5-7 days until discharge)
Time to readiness for extubation, time to extubation | Post ICU arrival POD 0 to discharge (2hours to on average 5-7 days until discharge)
Length of stay within ICU, readiness for discharge from the unit | Post ICU arrival POD 0 to discharge (2hours to on average 5-7 days until discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Wasowicz, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hopsital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Wasowicz M, Jerath A, Luksun W, Sharma V, Mitsakakis N, Meineri M, Katznelson R, Yau T, Rao V, Beattie WS. Comparison of propofol-based versus volatile-based anaesthesia and postoperative sedation in cardiac surgical patients: a prospective, randomized, study. Anaesthesiol Intensive Ther. 2018;50(3):200-209. doi: 10.5603/AIT.a2018.0012. Epub 2018 Jun 18. PMID 29913033
- [Derived] Pickworth T, Jerath A, DeVine R, Kherani N, Wasowicz M. The scavenging of volatile anesthetic agents in the cardiovascular intensive care unit environment: a technical report. Can J Anaesth. 2013 Jan;60(1):38-43. doi: 10.1007/s12630-012-9814-5. Epub 2012 Nov 7. PMID 23132045